CLINICAL TRIAL: NCT00023231
Title: Calcineurin Inhibitor Sparing Protocol in Living Donor Pediatric Kidney Transplantation
Brief Title: Pediatric Kidney Transplant Without Calcineurin Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CN01; CN01
Record Dates: First submitted 2001-08-29; First posted 2001-08-31 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Daclizumab; Methylprednisolone; Prednisone; Mycophenolic Acid; Sirolimus; Trimethoprim, Sulfamethoxazole Drug Combination; Ganciclovir; Atorvastatin

ARMS (1):
- 1 (Experimental): Participants will receive immunosuppression therapy using antibody induction (daclizumab), corticosteroids, mycophenolate mofetil, and sirolimus prior to transplantation. Bactrim and ganciclovir will be taken for infection prophylaxis. If the participant has consistent high levels of fasting cholesterol, treatment with lipitor may be given.
  Interventions: Drug: Daclizumab; Drug: Methylprednisolone/prednisone; Drug: Mycophenolate mofetil; Drug: Sirolimus; Drug: Bactrim; Drug: Ganciclovir; Drug: Lipitor

INTERVENTIONS:
Drug: Daclizumab — 1 mg/kg/dose at study entry and Weeks 2, 4, 6, and 8
  Other Names: Zenapax
Drug: Methylprednisolone/prednisone — Dosage is dependent on weight and varies throughout study. Refer to protocol for more information.
  Other Names: Cellcept
Drug: Mycophenolate mofetil — Solution or oral tablet taken daily. Dosage depends on body surface area.
Drug: Sirolimus — Oral tablet taken once prior to transplant. Dosage dependent on body surface area.
  Other Names: Rapamune
Drug: Bactrim — Oral tablet taken three times per week. Dosage is dependent on weight.
Drug: Ganciclovir — Oral tablet taken daily. Dosage is dependent on weight.
Drug: Lipitor — Oral tablet taken daily

SUMMARY:
The purpose of this study is to see the effect of using drugs other than calcineurin inhibitors to improve the rate of kidney transplant failure.

Kidney transplantation can help children with end-stage kidney disease. However, it has been difficult to find treatment for donor graft rejection that does not have a lot of side effects. Researchers hope to find treatments (immunosuppressants) with fewer side effects. One approach is to avoid using calcineurin inhibitors and to try a new drug known as sirolimus instead. Another is to use steroids less often. This study will test whether using sirolimus, fewer steroid treatments, MMF, and certain antibodies will improve long-term graft survival in children receiving kidney transplants from living donors.

DETAILED DESCRIPTION:
Renal transplantation is widely recognized as the treatment of choice for children with end-stage renal disease (ESRD). Although outcomes of renal transplantation in children have improved during the past decade, success has been limited by both non-specific tolerance and the complications associated with immunosuppressants. Steroids and calcineurin inhibitors have the most toxic side effects. Use of sirolimus for immunosuppression has not been associated with as many complications. Recent studies from Europe have demonstrated that sirolimus can be combined with MMF and steroids to provide excellent graft survival in the absence of calcineurin inhibitors. Steroid side-effects can be lessened by tapering the steroid dose to an every-other-day schedule. This protocol tests whether immunosuppression by IL-2r antibody, sirolimus, MMF, and alternate-day steroids will provide comparable graft survival for living donor recipients, compared to current immunosuppression, but with reduced complications of calcineurin inhibitors.

Evaluations prior to transplantation include a complete history and physical examination, CBC, liver function tests, and antibodies for CMV, EBV, HIV, HbsAG, and HCV. All appropriate vaccinations are provided before transplantation. Transplant recipients receive immunosuppression therapy using antibody induction (daclizumab), corticosteroids, mycophenolate mofetil, and sirolimus. Serum sirolimus levels are measured so that doses can be adjusted to maintain certain blood levels of the drug. Bactrim and ganciclovir are given for infection prophylaxis. If the patient has consistent high levels of fasting cholesterol, treatment with lipitor may be given. A transplant biopsy is performed at the time of the transplant and at 3, 6, and 12 months post transplantation and at times when a rejection is suspected. A radionuclide GFR is done at the same time points, and at 1, 24, and 36 months. The protocol biopsies, blood, and urine samples will be analyzed by genomic methods to determine differences in gene expression post transplantation. In the event of a first acute rejection, patients are treated with Solu-Medrol for 3 consecutive days. A second rejection (at the discretion of the transplant center) or severe rejection (Banff Grade 3) is treated with antibody therapy and, after a second or severe rejection, the immunosuppressant regimen is changed. Patients are followed for 36 months with routine physical examinations and laboratory assessments.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 21 years of age and under.
* Are kidney recipients of living-donor grafts, except when living-donor grafts are identically matched.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are recipients of identical (HLA matched) living-donor grafts.
* Are recipients of cadaver-donor grafts.
* Have certain abnormal kidney diseases that may return.
* Have failed 2 or more previous kidney transplants.
* Have fat abnormalities that are inherited or present at high levels.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2001-02; Primary Completion 2004-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment without calcineurin inhibitors, compared to current standard immunosuppressive treatment | Throughout study
Adverse effects of treatment without calcineurin inhibitors, compared to current standard immunosuppressive treatment, especially hypertension, serious infections and chronic nephrotoxicity | Throughout study

SECONDARY OUTCOMES:
Immune inhibition detected by sensitive and specific assays (including intragraft and peripheral monitoring) for expression patterns of activation and effector function markers | Throughout study

CONTACTS AND LOCATIONS:
Locations (1):
- Lauren Schenker, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Result] Harmon W, Meyers K, Ingelfinger J, McDonald R, McIntosh M, Ho M, Spaneas L, Palmer JA, Hawk M, Geehan C, Tinckam K, Hancock WW, Sayegh MH. Safety and efficacy of a calcineurin inhibitor avoidance regimen in pediatric renal transplantation. J Am Soc Nephrol. 2006 Jun;17(6):1735-45. doi: 10.1681/ASN.2006010049. Epub 2006 May 10. PMID 16687625
- [Result] Iacomini J, Sayegh MH. Measuring T cell alloreactivity to predict kidney transplant outcomes: are we there yet? J Am Soc Nephrol. 2006 Feb;17(2):328-30. doi: 10.1681/ASN.2005121264. Epub 2005 Dec 28. No abstract available. PMID 16382014
- [Result] Schachter AD, Meyers KE, Spaneas LD, Palmer JA, Salmanullah M, Baluarte J, Brayman KL, Harmon WE. Short sirolimus half-life in pediatric renal transplant recipients on a calcineurin inhibitor-free protocol. Pediatr Transplant. 2004 Apr;8(2):171-7. doi: 10.1046/j.1399-3046.2003.00148.x. PMID 15049798
- [Result] Hoerning A, Koss K, Datta D, Boneschansker L, Jones CN, Wong IY, Irimia D, Calzadilla K, Benitez F, Hoyer PF, Harmon WE, Briscoe DM. Subsets of human CD4(+) regulatory T cells express the peripheral homing receptor CXCR3. Eur J Immunol. 2011 Aug;41(8):2291-302. doi: 10.1002/eji.201041095. Epub 2011 Jun 24. PMID 21538345
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY131 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY131 — ImmPort study identifier is SDY131
- Available data/document: Study Protocol: SDY131 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY131 — ImmPort study identifier is SDY131
- Available data/document: Study summary, -design,-demographics, -mechanistic assays, -files et al.: SDY131 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY131 — ImmPort study identifier is SDY131